CLINICAL TRIAL: NCT03209154
Title: Individualized Blood Pressure Treatment: a Multidisciplinary Approach to Uncontrolled Hypertension in Order to Reduce Morbidity and Mortality
Brief Title: An Interventional Multidisciplinary Approach to Individualize Blood Pressure Treatment
Acronym: IDA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Sverre Erik Kjeldsen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017/6534
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Uncontrolled Hypertension
Keywords: Adherence; Therapeutic Drug Monitoring; Patient perspective
MeSH Terms: interventions — Drug Monitoring; Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Study Group intervention: Therapeutic drug monitoring.
  Interventions: Diagnostic Test: Therapeutic drug monitoring
- Control Group (Active Comparator): Control Group intervention: No intervention first 3 months. After 3 months of follow-up, half of the patients in the Control Group will be randomized to perform home blood pressure monitoring as an intervention. No intervention in the other half.
  Interventions: Device: Home blood pressure monitoring

INTERVENTIONS:
Diagnostic Test: Therapeutic drug monitoring — Therapeutic drug monitoring will be performed.
  Arms: Study Group
Device: Home blood pressure monitoring — Patients will perform home blood pressure monitoring at home.
  Arms: Control Group

SUMMARY:
The aim of the study is to investigate and explore the most important aspects of drug-adherence in the treatment of hypertension in order to improve treatment and blood pressure control, implying that new knowledge will reduce morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Uncontrolled hypertension
* A stable medication regimen for at least 4 weeks of ≥ 2 antihypertensive agents
* No planned changes in antihypertensive drugs

Exclusion Criteria:

* Withdrawal of consent
* 24-h systolic ambulatory blood pressure >/= 170 mmHg
* Patients with inadequate Norwegian language skills
* Positive pregnancy test
* Known alcohol or drug abuse
* estimated glomerular filtration rate <30 mL/min/1.73m2
* Albumin/creatinin ratio >300 mg/mmol
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | 3 months after baseline
  Change in systolic daytime ambulatory blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Sverre E Kjeldsen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Rognstad S, Soraas CL, Brunborg C, Halvorsen LV, Brobak KM, Olsen E, Bergland OU, Aune A, Tuv SS, Svarstad AC, Clasen PE, Haldsrud R, Larstorp ACK, Helland A, Opdal MS. Pharmacokinetic Variability of Amlodipine Serum Concentration and Effect on Blood Pressure in Patients Treated for Hypertension. Pharmacol Res Perspect. 2025 Aug;13(4):e70140. doi: 10.1002/prp2.70140. PMID 40616336
- [Derived] Halvorsen LV, Soraas CL, Larstorp ACK, Hjornholm U, Kjaer VN, Liestol K, Aune A, Olsen E, Brobak KM, Bergland OU, Rognstad S, Aarskog NR, Heimark S, Fadl Elmula FEM, Gerdts E, Mo R, Solbu MD, Opdal MS, Kjeldsen SE, Rostrup M, Hoieggen A. Effect of Therapeutic Drug Monitoring on Adherence and Blood Pressure: A Multicenter Randomized Clinical Trial. Am J Hypertens. 2024 Sep 16;37(10):826-836. doi: 10.1093/ajh/hpae059. PMID 38713475
- [Derived] Brobak KM, Halvorsen LV, Aass HCD, Soraas CL, Aune A, Olsen E, Bergland OU, Rognstad S, Blom KB, Birkeland JAK, Hoieggen A, Larstorp ACK, Solbu MD. Novel biomarkers in patients with uncontrolled hypertension with and without kidney damage. Blood Press. 2024 Dec;33(1):2323980. doi: 10.1080/08037051.2024.2323980. Epub 2024 Apr 12. PMID 38606688
- [Derived] Aune A, Ohldieck A, Halvorsen LV, Brobak KM, Olsen E, Rognstad S, Larstorp ACK, Soraas CL, Rossebo AB, Rosner A, Grytaas MA, Gerdts E. Gender Differences in Cardiac Organ Damage in Arterial Hypertension: Assessing the Role of Drug Nonadherence. High Blood Press Cardiovasc Prev. 2024 Mar;31(2):157-166. doi: 10.1007/s40292-024-00632-6. Epub 2024 Mar 26. PMID 38530572
- [Derived] Bergland OU, Halvorsen LV, Soraas CL, Hjornholm U, Kjaer VN, Rognstad S, Brobak KM, Aune A, Olsen E, Fauchald YM, Heimark S, Thorstensen CW, Liestol K, Solbu MD, Gerdts E, Mo R, Rostrup M, Kjeldsen SE, Hoieggen A, Opdal MS, Larstorp ACK, Fadl Elmula FEM. Detection of Nonadherence to Antihypertensive Treatment by Measurements of Serum Drug Concentrations. Hypertension. 2021 Sep;78(3):617-628. doi: 10.1161/HYPERTENSIONAHA.121.17514. Epub 2021 Jul 19. PMID 34275336